CLINICAL TRIAL: NCT01256164
Title: A U.S. Phase 2, Randomized, Single-Blind, Controlled, Comparative Efficacy and Safety Study of Topical Fibrocaps™ and Gelatin Sponge (USP) in Surgical Hemostasis
Brief Title: U.S. Study of Fibrocaps in Surgical Hemostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FC-002
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Hemorrhage
Keywords: fibrin sealants; hemostatics; time to hemostasis
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrocaps + Gelfoam (Experimental): After identification of a Target Bleeding Site (TBS), topical Fibrocaps should be applied using the Fibrospray device for general surgeries; and either the Fibrospray device or direct application for spinal and vascular surgeries, followed by application of Gelfoam and manual pressure with sterile gauze.
  Interventions: Device: Fibrocaps (fibrin sealant)
- Gelfoam (Active Comparator): Treatment is Gelfoam followed by manual pressure with sterile gauze. If hemostasis is not achieved within 10 minutes of the Start Time,the subject should be considered a treatment failure and the surgeon should implement additional hemostatic measures.
  Interventions: Device: Gelfoam

INTERVENTIONS:
Device: Fibrocaps (fibrin sealant) — Fibrocaps powder (max dose 1.5g) should be applied directly to the bleeding site or to the Gelfoam and then applied to the bleeding site. Re-application of 1.5 g of Fibrocaps is allowed.
  Other Names: Pro-0601
  Arms: Fibrocaps + Gelfoam
Device: Gelfoam — An identified Target Bleeding Site (TBS) should be treated with application of Gelfoam followed by light manual pressure with a sterile gauze.
  Arms: Gelfoam

SUMMARY:
The purpose of this study was to characterize the safety and hemostatic activity of topical Fibrocaps in surgical patients when control of mild to moderate bleeding by standard surgical techniques was ineffective and/or impractical.

DETAILED DESCRIPTION:
This was a multi-center, prospective, randomized, single-blind, controlled, comparative efficacy and safety trial in 90 subjects undergoing spinal surgery, hepatic resection, specific soft tissue dissection, or peripheral vascular surgery, ((including peripheral artery bypass and arteriovenous graft formation for hemodialysis using either Polytetrafluoroethylene (PTFE) or native grafts)). Subjects were randomized in a 2:1 ratio to Fibrocaps + Gelfoam or Gelfoam on the day of surgery.

Use of the Fibrospray device was optional for spinal and vascular surgeries, but required for the general surgery procedures. All investigators using the Fibrospray device were trained on the correct and safe set-up and use of Fibrocaps and the Fibrospray device prior to participating in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 years of age or older
* Subjects who are able and willing to provide written and signed informed consent
* All subjects willing to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits
* A life expectancy of at least one year

Intra-Operative inclusion criteria

* Presence of mild or moderate bleeding/oozing when control by conventional surgical techniques, including but not limited to suture, ligature and cautery is ineffective or impractical
* Absence of intraoperative complications other than bleeding which, in the opinion of the investigator, may interfere with the assessment of efficacy or safety
* No intraoperative use of a topical hemostat containing thrombin
* Approximate Target Bleeding Site surface area of no more than 100 square centimeters

Exclusion Criteria:

* Pregnant or lactating women
* Has a known intolerance to blood products or to Fibrocaps components
* Unwilling to receive human blood products
* Subject has a known allergy to porcine gelatin
* Has a mental or physical condition that would, in the opinion of the investigator, place the subject at an unacceptable risk or render the subject unable to meet the requirements of the protocol
* Currently participating or has participated in another clinical study involving another investigational agent within 4 weeks of the start of this trial, or is planning participation in another clinical trial during the 4 weeks after surgery
* Has any clinically-significant coagulation disorder that may interfere with the assessment of efficacy or pose a safety risk to the subject according to the investigator
* Aspartate Aminotransferase (AST) or Alanine aminotransferase (ALT) 3 times (or more) the upper limit normal range during screening, except for subjects undergoing liver resection surgery where there is no upper limit for these analytes due to the nature of their disease.
* Platelets < 10 x 10^9 /L during screening
* Activated partial thromboplastin time (aPTT) > 100 seconds during screening
* International normalized ratio (INR)greater than 2.5 during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Frohna, MD, PhD, Study Director — Mallinckrodt
Locations (1):
- Various sites, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in February 2011 and completed in October 2011 at 8 investigative study sites in the United States.
Pre-assignment Details: Approximately 90 eligible subjects were planned for enrollment, randomization, and treatment. The enrollment stopped short of the targeted 90 subjects due to enrollment of more subjects in the parallel study being conducted in the Netherlands.
Groups:
- Fibrocaps + Gelfoam: After identification of a Target Bleeding Site (TBS), topical Fibrocaps powder will be applied using the Fibrospray device for general surgeries; and either the Fibrospray device or direct application for spinal and vascular surgeries, followed by application of Gelfoam and manual pressure with sterile gauze.
- Gelfoam: Treatment will be Gelfoam followed by manual pressure with sterile gauze. If hemostasis has not been achieved within 10 minutes of the Start Time,the subject will be considered a treatment failure and the surgeon will implement additional hemostatic measures.
Period: Overall Study
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Started | 47 | 23
Completed | 47 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrocaps + Gelfoam | Gelfoam | Total
Number analyzed (Participants) | 47 | 23 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 13 | 39
  >=65 years | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (13.97) | 61.3 (10.48) | 59.8 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 14 | 36
  Male | 25 | 9 | 34
Region of Enrollment [Number; unit: participants]
  United States | 47 | 23 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Hemostasis (TTH)
Description: Time to hemostasis recorded from the first application of study treatment until cessation of bleeding
Time Frame: 0-10 minutes
Population: All subjects treated with a time to hemostasis were included in the analysis
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Number analyzed (Participants) | 47 | 23
minutes | 1.9 (1.3) | 4.8 (3.1)
Statistical Analysis 1: Comparison: Fibrocaps + Gelfoam vs Gelfoam; Test type: Non-Inferiority or Equivalence — With 90 subjects, randomized on a 2:1 ratio into the Fibrocaps plus gelatin sponge active arm or the gelatin sponge arm, and assuming a mean TTH of 3.5 minutes with a standard deviation of 2.5 minutes in the active arm and a mean TTH of 6 minutes in the control arm, this translates in a power of 99.4% at a two-sided significance level alpha of 5%, using a two-sample t-test; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Safety
Description: Number of participants with Adverse events and clinically-significant changes/findings on labs and physical examination as well as incidence of re-operation for bleeding at the TBS
Time Frame: 28 Days
Population: All subjects treated were analyzed for safety.
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Number analyzed (Participants) | 47 | 23
participants | 47 | 23
Statistical Analysis 1: Comparison: Fibrocaps + Gelfoam vs Gelfoam; Test type: Superiority or Other; p = 1.00, t-test, 2 sided

3. Secondary Outcome: Number of Subjects Achieving Hemostasis at 3 Minutes
Time Frame: 3 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Number analyzed (Participants) | 47 | 23
participants | 39 | 8
Statistical Analysis 1: Comparison: Fibrocaps + Gelfoam vs Gelfoam; Intent-to-treat analysis; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Number of Participants Achieving Hemostasis at 5 Minutes
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Number analyzed (Participants) | 47 | 23
participants | 44 | 14
Statistical Analysis 1: Comparison: Fibrocaps + Gelfoam vs Gelfoam; intent-to- treat analysis; Test type: Superiority or Other; p = 0.001, Fisher Exact

5. Secondary Outcome: Number of Patients Achieving Hemostasis at 10 Minutes
Time Frame: 10 minutes
Measure: Number; unit: participants
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Number analyzed (Participants) | 47 | 23
participants | 47 | 18
Statistical Analysis 1: Comparison: Fibrocaps + Gelfoam vs Gelfoam; intent-to-treat analysis; Test type: Superiority or Other; p = 0.003, Fisher Exact

ADVERSE EVENTS:
Time Frame: Treatment emergent Adverse Events (AE) were collected for 28 days post treatment
Arm/Group | Fibrocaps + Gelfoam | Gelfoam
Serious Adverse Events (participants affected / at risk) | 6/47 | 2/23
Other Adverse Events (participants affected / at risk) | 44/47 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrocaps + Gelfoam (N=47) | Gelfoam (N=23)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary emobolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep cenous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Scrotal hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibrocaps + Gelfoam (N=47) | Gelfoam (N=23)
Constipation (Gastrointestinal disorders) | 12 (12) | 5 (5)
Nausea (Gastrointestinal disorders) | 15 (15) | 9 (9)
Vomiting (Gastrointestinal disorders) | 8 (8) | 2 (2)
Oedema peripheral (General disorders) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Incision site pain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 25 (25) | 12 (12)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (26)
Headache (Nervous system disorders) | 6 (6) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators were part of the primary publication. Each investigator may publish on the data from subjects enrolled at their site after the initial publication has been submitted.